CLINICAL TRIAL: NCT02616640
Title: A Phase IB Multicenter, Open-label Study To Determine The Recommended Dose And Regimen Of Durvalumab (MEDI4736) Either As Monotherapy or In Combination With Pomalidomide (POM) With Or Without Low-Dose Dexamethasone (DEX) In Subjects With Relapsed And Refractory Multiple Myeloma (RRMM)
Brief Title: A Study to Determine Dose and Regimen of Durvalumab as Monotherapy or in Combination With Pomalidomide With or Without Dexamethasone in Subjects With Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MEDI4736-MM-001
Record Dates: First submitted 2015-11-25; First posted 2015-11-30 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Relapsed; Refractory; MEDI4736; Durvalumab; Pomalidomide (POM); Dexamethasone (DEX); PD-L1
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — durvalumab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Durvalumab monotherapy (Experimental): Intravenous (IV) durvalumab at assigned dose level (750, 1500, 2250, or 3000 mg) over 1 hour on day 1 of a 28-day cycle
  Interventions: Drug: Durvalumab
- Durvalumab + pomalidomide (POM) (Experimental): IV durvalumab at assigned dose level (750, 1500, 2250, or 3000 mg) over 1 hour on day 1 of a 28-day cycle and Oral POM 4 mg/day on Days 1 to 21 of each 28-day treatment cycle
  Interventions: Drug: Durvalumab; Drug: Pomalidomide
- Durvalumab + pomalidomide (POM) + dexamethasone (dex) (Experimental): IV durvalumab at assigned dose level (750, 1500, 2250, or 3000 mg) over 1 hour on day 1 of a 28-day cycle with Oral POM 4 mg/day on Days 1 to 21 of each 28-day treatment cycle and Oral dex 40 mg/day (≤ 75 years old) or 20 mg/day (> 75 years old) on Days 1, 8, 15, and 22 of a 28-day cycle
  Interventions: Drug: Durvalumab; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Durvalumab
  Other Names: MEDI4736
Drug: Pomalidomide
  Arms: Durvalumab + pomalidomide (POM); Durvalumab + pomalidomide (POM) + dexamethasone (dex)
Drug: Dexamethasone
  Arms: Durvalumab + pomalidomide (POM) + dexamethasone (dex)

SUMMARY:
This is a multicenter, open-label, Phase 1b study to determine the recommended dose and regimen of durvalumab either as monotherapy or in combination with POM with or without low dose dex in subjects with RRMM. The study will consist of a dose-finding portion as well as a parallel dose-expansion portion to determine the optimal dose and regimen.

On 05 Sep 2017, a Partial Clinical Hold was placed on this study by the United States (US) Food and Drug Administration (FDA). The decision by the FDA was based on data related to risks of anti-programmed cell death-1 (PD-1) antibody, pembrolizumab, in combination with IMiDs® immunomodulatory drugs in patients with multiple myeloma. As a result, enrollment into this study has been discontinued. Subjects who are receiving clinical benefit, based on the discretion of the investigator, may remain on study treatment after being reconsented.

ELIGIBILITY:
Inclusion Criteria:

* Has a confirmed diagnosis of active multiple myeloma and measurable disease.
* Must have undergone prior treatment with ≥2 treatment lines of anti-myeloma therapy
* Must have failed last line of treatment (refractory to last line of treatment).
* Must have achieved at least a stable disease (SD) for at least 1 cycle of treatment to at least 1 prior anti-myeloma regimen before developing Progressive disease (PD) (relapsed)
* Prior anti-myeloma treatments must have included a lenalidomide AND proteasome inhibitor alone or in combination.
* Has performance status of 0, 1, or 2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
* The extramedullary plasmacytoma (EMP) sub-group, must have radiologically measurable EMP disease (soft tissue or bone related) that is amenable to biopsy and does not need to have measurable disease.

Exclusion Criteria:

* Has non-secretory or oligosecretory multiple myeloma
* Has had prior anti-myeloma therapy within 2 weeks prior to study Day 1
* Has undergone prior organ or allogeneic hematopoetic stem cell transplantation
* Has received previous therapy with pomalidomide and did not achieve at least a stable disease
* Has received prior therapy with an anti-programmed cell death 1 receptor (anti-PD-1), antiprogrammed death-ligand 1 (anti-PD-L1), antiprogrammed death-ligand 2 (anti-PD-L2), anti-CD137, or anti-cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell costimulation or checkpoint pathways).
* Has received prior treatment with a monoclonal antibody within 5 half-lives of Study Day 1
* Has received investigational agents within 28 days or 5 half-lives (whichever is longer) of Study Day 1
* Has received live, attenuated vaccine within 30 days prior to Study Day 1
* Had rash ≥ Grade 3 during prior thalidomide, lenalidomide, or pomalidomide therapy
* Has a history of anaphylaxis or hypersensitivity to thalidomide, lenalidomide, POM, or dex
* Has peripheral neuropathy ≥ Grade 2
* Has a known additional malignancy that is progressing or requires active treatment (except for basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy).
* Is positive for human immunodeficiency virus (HIV), chronic or active hepatitis B or active hepatitis A or C
* Has a prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 5 years (with the exception Basal cell carcinoma of the skin, Squamous cell carcinoma of the skin, Carcinoma in situ of the cervix, Carcinoma in situ of the breast, Incidental histologic finding of prostate cancer [T1a or T1b] or prostate cancer that is curative)
* Has clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS multiple myeloma
* Has clinically significant cardiac disease
* Is a female who is pregnant, nursing, or breastfeeding, or who intends to become pregnant during the participation in the study
* Is a current smoker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2018-11-23 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Dose-limiting Toxicities (DLTs) | Approximately 1 month
  Number of participants with DLTs in the first cycle of treatment

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to approximately 2 year
  Number of participants with adverse events
Overall response rate (ORR) | Up to approximately 2 year
  Tumor response, including progressive disease (PD) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria
Time to response (TTR) | Up to approximately 2 year
  Time from first dose to the first documentation of response (Partial Response [PR] or greater)
Duration of response (DOR) | Up to approximately 2 year
  Is defined as time from the earliest date of documented response (partial response (PR) or better) to the earliest date when disease progression was confirmed
Pharmacokinetics- Cmax | Up to approximately 1 year
  Maximum observed concentration
Pharmacokinetics- AUC | Up to approximately 1 year
  Area under the concentration-time curve
Pharmacokinetics- Tmax | Up to approximately 1 year
  Time to maximum concentration
Pharmacokinetics- t1/2 | Up to approximately 1 year
  Terminal elimination half-life
Pharmacokinetics- CL/F | Up to approximately 1 year
  Apparent total body clearance
Pharmacokinetics- Vz/F | Up to approximately 1 year
  Volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Lars Sternas, MD, PhD, Study Director — Celgene Corporation
Locations (22):
- United States (8):
  - Local Institution - 102, Baltimore, Maryland
  - Local Institution - 114, Boston, Massachusetts
  - Local Institution - 108, Boston, Massachusetts
  - Local Institution - 115, Boston, Massachusetts
  - Local Institution - 105, New York, New York
  - Local Institution - 106, Charlotte, North Carolina
  - Local Institution - 110, Cleveland, Ohio
  - Local Institution - 107, Milwaukee, Wisconsin
- Local Institution - 201, Calgary, Alberta, Canada
- France (3):
  - Local Institution - 601, Lille
  - Local Institution - 602, Poitiers
  - Local Institution - 603, Toulouse
- Local Institution - 301, Tübingen, Germany
- Italy (3):
  - Local Institution - 403, Pavia
  - Local Institution - 405, Rozzano (MI)
  - Local Institution - 401, Torino
- Netherlands (2):
  - Local Institution - 702, Amsterdam
  - Local Institution - 701, Rotterdam
- Spain (4):
  - Local Institution - 501, Barcelona
  - Local Institution - 504, Madrid
  - Local Institution - 502, Pamplona
  - Local Institution - 505, Valencia

REFERENCES:
- [Derived] Young MH, Pietz G, Whalen E, Copeland W, Thompson E, Fox BA, Newhall KJ. Immunomodulation by durvalumab and pomalidomide in patients with relapsed/refractory multiple myeloma. Sci Rep. 2021 Aug 12;11(1):16460. doi: 10.1038/s41598-021-95902-x. PMID 34385543
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/home